CLINICAL TRIAL: NCT06351449
Title: Characterization of Visual Characteristics in Allergic Contact Dermatitis Using the Skincam® Tool
Acronym: PatchCam
Status: Not yet recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL22_0489
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Allergic Contact Dermatitis
Keywords: Allergic contact dermatis (ACD); Patch Test; Photographs; SkinCams
MeSH Terms: conditions — Dermatitis, Allergic Contact

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with allergic contact dermatitis history: Adult patients with allergic contact dermatitis history and requiring patch test during their care pathway and accepting unidentified photographs of patch test results.
  Interventions: Other: The patch under study is photographed using the SkinCam®

INTERVENTIONS:
Other: The patch under study is photographed using the SkinCam® — Unlike standard care, the patch under study is photographed using the SkinCam® and not a standard camera. The shooting and photographic remain similar to that of standard care, with only the camera used being changed.

SUMMARY:
Contact dermatitis (CD) is a common inflammatory skin disease, affecting approximately 15-20% of the general population in industrialized countries and ranking first among occupational diseases in many European countries.

The patch test method aims at reproducing the eczematous lesions by applying occlusive patches containing the suspected allergens to the patient's healthy skin. It requires experienced medical staff to read the reaction.

Newtones Technologies society has developed a new tool, the SkinCam®, able to capture high resolution cross and parallel images, allowing a quantification of color and relief of skin.

This study aims to illustrate patch test results, describing skin appearance (color, roughness, shine), using photographs taken by the SkinCam®.

DETAILED DESCRIPTION:
Contact dermatitis (CD) is a common inflammatory skin disease, affecting approximately 15-20% of the general population in industrialized countries and ranking first among occupational diseases in many European countries.

Allergic contact dermatitis (ACD) typically presents as a severe skin inflammation with redness, edema, oozing and crusting. It is characterized by a delayed type IV hypersensitivity response mediated by allergen-specific T cells in sensitized individuals. Current diagnosis relies on clinical investigations by diagnostic patch testing with suspected allergenic chemicals.

The patch test method aims at reproducing the eczematous lesions by applying occlusive patches containing the suspected allergens to the patient's healthy skin. It requires experienced medical staff to read the reaction.

Newtones Technologies society has developed a new tool, the SkinCam®, able to capture high resolution cross and parallel images, allowing a quantification of color and relief of skin.

This study aims to illustrate patch test results, describing skin appearance (color, roughness, shine), using photographs taken by the SkinCam®.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, over 18 years of age
* Patients called for reading patch test, applied 72 or 96 hours ago
* Patients agreeing to have unidentified photographs of patchs tests
* Patient affiliated to or benefiting from a social security regime
* Patient having been informed and not having opposed

Exclusion Criteria:

* Protected patient: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision
* Pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for suspected contact dermatitis to the Allergology and Clinical Immunology Department of the Centre Hospitalier Lyon Sud and the Dermatology and Allergology Department of the Centre Hospitalier Universitaire de St Etienne, with allergic contact dermatitis history and requiring patch test during their care pathway
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-04-15 (Estimated); Primary Completion 2027-04-15 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
To highlight characteristics of allergic contact dermatitis (ACD) | one day
  To highlight characteristics of allergic contact dermatitis (ACD), illustrating visually positive patch tests (+, ++, +++) with numerical parameters (colorimetry, shine and roughness)